CLINICAL TRIAL: NCT01528280
Title: Vaccination Against Hepatitis A Virus in Shift Workers: Evaluation of the Humoral and Cellular Immune Response
Brief Title: Humoral and Cellular Response in Shift Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marco Tulio de Mello, Associate Professor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CEPE2012FRuiz
Record Dates: First submitted 2012-02-02; First posted 2012-02-08 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Other Condition That May be a Focus of Clinical Attention
Keywords: Shift work; Hepatitis A vaccination; humoral response; cellular response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Shiftwork (Experimental): The comparison will consider nightworkers versus dayworkers.
  Interventions: Biological: Vaccination against hepatitis A; Other: No Intervention

INTERVENTIONS:
Biological: Vaccination against hepatitis A — Vaccination against hepatitis A (2 doses) into the deltoid muscle of the nondominant arm twice, i.e., at 0 and 6 months.
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to access whether shift workers (morning, afternoon or night) vaccinated against hepatitis A would have some humoral and cellular response impairment.

DETAILED DESCRIPTION:
Sleep regulates immune functions. In this sense, we asked whether shift workers (morning, afternoon or night) vaccinated against hepatitis A would have some humoral and cellular response impairment. Men (18 to 55 years) will be recruited through different forms of media (electronic, newspapers, radio and magazines). The shift workers sleep pattern will be recorded polysomnographically. Subsequently, the volunteers will be underwent vaccination against hepatitis A (2 doses) and after 30, 60 and 90 days, blood samples will be collected to assess the humoral response in the experimental groups. The hormones prolactin, growth hormone, cortisol, adrenaline and noradrenaline will also be evaluated. Indeed, stimulations in culture will be conducted to assess the cellular response profile against the vaccination through the production assessment of IL-4, IFN-γ, IL-2 and TNF-α.

ELIGIBILITY:
Inclusion Criteria:

* shift workers
* naive immune status against hepatitis A confirmed by hepatitis A virus (HAV) antibodies levels below 5 mIU/mL

Exclusion Criteria:

* smokers
* individuals with complaints and/or sleep disorders
* acute or chronic disease
* use of medication during the study period.
* acute illnesses

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Antibodies against hepatitis A virus (anti-HAV) | Baseline, 30 days, 60 days and 90 days
  Change in antibodies against hepatitis A virus (anti-HAV) production

SECONDARY OUTCOMES:
Intracellular cytokines | Baseline, 30 days, 60 days and 90 days
  Change in intracellular IL-4, IFN-γ, IL-2 e TNF-α cytokine levels
Catecholamines | Baseline, 30 days, 60 days and 90 days
  Change in cathecolamines levels
Prolactin | Baseline, 30 days, 60 days and 90 days
  Change in prolactin levels
Growth hormone | Baseline, 30 days, 60 days and 90 days
  Change in growth hormone levels
Cortisol | Baseline, 30 days, 60 days and 90 days
  Change in cortisol levels
Sleep disorders | Baseline
  Assessment of sleep disorders

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tulio Mello, Associate Professor, Study Director — Federal University of São Paulo; Francieli Silva Ruiz, PhD, Study Chair — Federal University of São Paulo; Andrea Maculano, PhD, Study Chair — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - Centro de Estudos em Psicobiologia e Exercicio _ CEPE, São Paulo, São Paulo
  - Centro de Estudos em Psicobiologia e Exercicio - CEPE, São Paulo

REFERENCES:
- See also: Fundação de Amparo à Pesquisa do Estado de São Paulo — http://www.fapesp.br/